CLINICAL TRIAL: NCT02227446
Title: Local Antibiotic Therapy to Reduce Infection After Operative Treatment of Fractures at High Risk of Infection: A Multicenter Randomized, Controlled Trial (Vancomycin Study)
Brief Title: Local Antibiotic Therapy to Reduce Infection After Operative Treatment of Fractures at High Risk of Infection: A Multicenter Randomized, Controlled Trial (VANCO)
Acronym: VANCO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Major Extremity Trauma Research Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH-10-2-0134
Record Dates: First submitted 2014-08-21; First posted 2014-08-28 (Estimated); Results first posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Post Operative Surgical Site Infection
Keywords: Surgical site infection risk prevention; Bacterial species type and antibacterial sensitives

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vancomycin Antibotic Powder (Experimental): Participants in the treatment group will receive the study intervention of a maximum dose of 1000mg of Vancomycin antibiotic powder in their wound bed, which is placed right before wound closure. Vancomycin antibiotic powder may be combined with normal saline as per clinical practice at the participating institution.
  In addition, participants in this group will receive standard of care treatment for their injury, to include all institution specific standard treatment (prophylactic and otherwise) for preventing and treating infection.
  Interventions: Drug: Vancomycin antibiotic powder
- Standard of Care (No Intervention): Participants in this group will receive standard of care treatment for their injury, to include all institution specific standard treatment (prophylactic and otherwise) for preventing and treating infection. Participants in this group will not receive local Vancomycin antibiotic powder.

INTERVENTIONS:
Drug: Vancomycin antibiotic powder — At the time of fracture fixation 1000 mg of Vancomycin powder placed into the wound during wound closure.
  Arms: Vancomycin Antibotic Powder

SUMMARY:
The Vancomycin Study is a multi-center, prospective randomized controlled trial that will compare the proportion of deep surgical site infections within 6 months in patients treated with local Vancomycin powder compared to those treated without local Vancomycin powder at the time of fracture fixation.

DETAILED DESCRIPTION:
Primary Aim: Compare the proportion of deep surgical site infections within 6 months in patients treated with local Vancomycin powder compared to those treated without local Vancomycin powder.

Primary Hypothesis: The proportion of deep surgical site infections will be lower for patients treated with local Vancomycin powder.

Secondary Aim #1: Compare antibiotic sensitivities of the bacteria in the patients who develop deep surgical site infections in study patients treated with local Vancomycin powder compared to those treated without local Vancomycin powder.

Hypothesis 1: In the patients who develop infections, the antibiotic sensitivity profiles between patients treated with local Vancomycin powder will be non-inferior to those treated without local Vancomycin powder.

Secondary Aim #2: Build and validate a risk prediction model for the development of deep surgical site infections in patients treated without local Vancomycin powder. (b) Explore whether the effect of local Vancomycin powder is modified by the predicted risk of infection.

Hypothesis 2: Patient (e.g. medical co-morbidities) and injury (e.g open fractures) factors will be highly predictive of infection risk.

Hypothesis 3: Patients with higher predictive risk will experience greater benefit from local antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* All "high energy" tibial plateau fractures treated operatively with plate and screw fixation.
* We define "high energy" tibial plateau fractures as patients who are either:

  * Initially treated with an external fixation (with or without limited internal fixation) and treated definitively more than 3 days later after swelling has resolved.
  * Any open type I, II, or IIIA fracture, regardless of timing of definitive treatment.
  * Any tibial plateau fracture associated with ipsilateral leg compartment syndrome fasciotomy wounds.
* All "high energy" pilon (distal tibial plafond) fractures treated operatively with plate and screw fixation. We define "high energy" pilon fractures as patients who are either:

  * Initially treated with an external fixation (with or without fibula fixation or limited internal fixation) and treated definitively more than 3 days later after swelling has resolved.
  * Any open type I, II, or IIIA fracture, regardless of timing of definitive treatment.
  * Any tibial pilon fracture associated with ipsilateral leg compartment syndrome fasciotomy wounds.
* Ages 18 to 80 years
* Patients may have co-existing non-tibial infection, with or without antibiotic treatment.
* Patients may have risk factors for infection including diabetes, immunosuppression from steroids or other medications, HIV, or other infections.
* Patients may have a head injury
* Patients may have a portion of the fixation (e.g. fibula fixation in pilon or percutaneous screws across a tibial plateau fracture) prior to definitive plate fixation, at the initial surgery before randomization.
* Patients may have other orthopedic and non-orthopaedic injuries.
* Patients may have pre-existing musculoskeletal injuries, be non ambulators, or have spinal cord injuries.
* Women and minorities are included

Exclusion Criteria:

* The study injury: tibial plateau, pilon, is already infected at time of study enrollment.
* Patient speaks neither English nor Spanish.
* Patients who have already had definitive fixation prior to enrollment in the study.
* Severe problems with maintaining follow-up (e.g. patients who are homeless at the time of injury or those how are intellectually challenged without adequate family support).
* Patients with allergies, drug administration reactions, or other sensitivities to Vancomycin (such as a history of Redman's Syndrome).
* Pregnancy.
* The study injury is a type IIIB or IIIC open fracture.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1036 (Actual)
Dates: Start 2014-10; Primary Completion 2018-06 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renan Castillo, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Robert O'Toole, MD, Principal Investigator — University of Maryland R Adams Cowley Shock Trauma Center; Anthony Carlini, MS, Study Director — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- University of Maryland R Adams Cowley Shock Trauma Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Major Extremity Trauma Research Consortium (METRC); O'Toole RV, Joshi M, Carlini AR, Murray CK, Allen LE, Huang Y, Scharfstein DO, O'Hara NN, Gary JL, Bosse MJ, Castillo RC, Bishop JA, Weaver MJ, Firoozabadi R, Hsu JR, Karunakar MA, Seymour RB, Sims SH, Churchill C, Brennan ML, Gonzales G, Reilly RM, Zura RD, Howes CR, Mir HR, Wagstrom EA, Westberg J, Gaski GE, Kempton LB, Natoli RM, Sorkin AT, Virkus WW, Hill LC, Hymes RA, Holzman M, Malekzadeh AS, Schulman JE, Ramsey L, Cuff JAN, Haaser S, Osgood GM, Shafiq B, Laljani V, Lee OC, Krause PC, Rowe CJ, Hilliard CL, Morandi MM, Mullins A, Achor TS, Choo AM, Munz JW, Boutte SJ, Vallier HA, Breslin MA, Frisch HM, Kaufman AM, Large TM, LeCroy CM, Riggsbee C, Smith CS, Crickard CV, Phieffer LS, Sheridan E, Jones CB, Sietsema DL, Reid JS, Ringenbach K, Hayda R, Evans AR, Crisco MJ, Rivera JC, Osborn PM, Kimmel J, Stawicki SP, Nwachuku CO, Wojda TR, Rehman S, Donnelly JM, Caroom C, Jenkins MD, Boulton CL, Costales TG, LeBrun CT, Manson TT, Mascarenhas DC, Nascone JW, Pollak AN, Sciadini MF, Slobogean GP, Berger PZ, Connelly DW, Degani Y, Howe AL, Marinos DP, Montalvo RN, Reahl GB, Schoonover CD, Schroder LK, Vang S, Bergin PF, Graves ML, Russell GV, Spitler CA, Hydrick JM, Teague D, Ertl W, Hickerson LE, Moloney GB, Weinlein JC, Zelle BA, Agarwal A, Karia RA, Sathy AK, Au B, Maroto M, Sanders D, Higgins TF, Haller JM, Rothberg DL, Weiss DB, Yarboro SR, McVey ED, Lester-Ballard V, Goodspeed D, Lang GJ, Whiting PS, Siy AB, Obremskey WT, Jahangir AA, Attum B, Burgos EJ, Molina CS, Rodriguez-Buitrago A, Gajari V, Trochez KM, Halvorson JJ, Miller AN, Goodman JB, Holden MB, McAndrew CM, Gardner MJ, Ricci WM, Spraggs-Hughes A, Collins SC, Taylor TJ, Zadnik M. Effect of Intrawound Vancomycin Powder in Operatively Treated High-risk Tibia Fractures: A Randomized Clinical Trial. JAMA Surg. 2021 May 1;156(5):e207259. doi: 10.1001/jamasurg.2020.7259. Epub 2021 May 12. PMID 33760010
- See also: Related Info — http://metrc.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 1000 participants (500 per treatment arm) were enrolled across 36 METRC trauma centers over a 30-month period. Participants were recruited during the initial hospitalization for the their injury.
Groups:
- Control: Participants randomized to the control arm received standard infection prevention protocol without 1000 mg of intrawound vancomycin powder.
- Vancomycin Powder: Participants randomized to the intervention arm received standard infection prevention protocol with 1000 mg of intrawound vancomycin powder.
Period: Overall Study
Arm/Group | Control | Vancomycin Powder
Started | 521 | 515
Completed | 499 | 481
Not Completed | 22 | 34
Not completed — not eligible post randomization | 18 | 29
Not completed — Withdrawal by Subject | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Vancomycin Antibiotic Powder: Participants in the treatment group will receive the study intervention of a maximum dose of 1000mg of Vancomycin antibiotic powder in their wound bed, which is placed right before wound closure. Vancomycin antibiotic powder may be combined with normal saline as per clinical practice at the participating institution.
  In addition, participants in this group will receive standard of care treatment for their injury, to include all institution specific standard treatment (prophylactic and otherwise) for preventing and treating infection.
  Vancomycin antibiotic powder: At the time of fracture fixation 1000 mg of Vancomycin powder placed into the wound during wound closure.
- Total: Total of all reporting groups
Arm/Group | Vancomycin Antibiotic Powder | Standard of Care | Total
Number analyzed (Participants) | 481 | 499 | 980
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age (SD) in each study arm. Population: Numbers differ because each arm had a different number of participants.
  years | 45.4 (14) | 46.1 (13.5) | 45.75 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 181 | 363
  Male | 299 | 318 | 617
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 49 | 58 | 107
  Non-Hispanic White | 339 | 346 | 685
  Non-Hispanic Black | 71 | 77 | 148
  Other | 19 | 15 | 34
  Refused/Unknown | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Clinically Significant Deep Surgical Site Infection (SSI)
Description: The main outcome will be the presence of clinically significant surgical site infection (SSI) in the first 26 weeks after surgery, as determined by CDC guidelines. The CDC criteria is currently 3 months for surgical site infection. To help capture more infections the study investigators have moved the time frame back to 6 months.
  Wound characteristics will also be evaluated using the ASEPSIS score. In this system wounds are scored using the weighted sum of points assigned for predetermined criteria including the need for Additional treatment, presence of Serous drainage, Erythema, Purulent exudates, Separation of deep tissues, the Isolation of bacteria, and the duration of patients Stay (ASEPSIS).
  The study investigators will define deep infections as those that require operative treatment, and superficial infections as those that are treated without operative intervention.
Time Frame: 26 weeks
Measure: Count of Units; unit: surgical site infections
Units Other Than Participants: surgical site infections
Groups:
- Vancomycin Antibotic Powder: Participants in the treatment group will receive the study intervention of a maximum dose of 1000mg of Vancomycin antibiotic powder in their wound bed, which is placed right before wound closure. Vancomycin antibiotic powder may be combined with normal saline as per clinical practice at the participating institution.
  In addition, participants in this group will receive standard of care treatment for their injury, to include all institution specific standard treatment (prophylactic and otherwise) for preventing and treating infection.
  Vancomycin antibiotic powder: At the time of fracture fixation 1000 mg of Vancomycin powder placed into the wound during wound closure.
Arm/Group | Vancomycin Antibotic Powder | Standard of Care
Number analyzed (Participants) | 481 | 499
Number analyzed (surgical site infections) | 481 | 499
surgical site infections
  Total deep Surgical Site Infections | 29 | 48
  Culture negative deep SSI | 1 | 1
  Gram positive deep SSI | 17 | 36
  Gram negative deep SSI | 11 | 10
  Anerobe/fungal deep SSI | 1 | 0
  Contaminated sample | 0 | 1

2. Secondary Outcome: Bacterial Antibiotic Resistance Rate of Infected Participants
Description: Secondary outcome measures in this study include culture data in the group that becomes infected. Sensitivities of the isolate determined routinely in current clinical practice, will be recorded for analysis.
  The most common bacterial isolates in infection after orthopaedic fracture care are methicillin resistant staph. aureus and methicillin resistant coagulase negative Staphylococci. The rate of bacterial Vancomycin sensitivity will be measured and analyzed.
Time Frame: 26 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Identify Risk Factors for Infection
Description: A secondary outcome measure will be to determine the risk for postoperative infection as well as determine which patients are most likely to benefit from the local Vancomycin powder technique.
  Demographic variables will include age, presence of co-morbidities such as diabetes, smoking history, history of prior musculoskeletal infection, and history of infection within the past 30 days.
  Injury descriptors will include injury mechanism, open or closed fracture type, AO classification of the fracture type, other orthopaedic injuries, and other non-orthopaedic injuries.
  Treatment parameters will include time from injury to definitive treatment, time from injury to external fixation, and surgical approaches used.
Time Frame: 26 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | Control | Vancomycin Powder
All-Cause Mortality (participants affected / at risk) | 3/499 | 4/481
Serious Adverse Events (participants affected / at risk) | 21/499 | 16/481
Other Adverse Events (participants affected / at risk) | 0/499 | 0/481
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=499) | Vancomycin Powder (N=481)
Infection (Infections and infestations) | 6 (6) | 3 (3)
Abdominal injury (Gastrointestinal disorders) | 1 (1) | 5 (5)
Venous thromboembolism (VTE) (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Nonunion (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Manipulation under anesthesia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Amputation (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Hip fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Abnormal laboratory values (General disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Reaction to antibiotic (General disorders) | 1 (1) | 0 (0)
Renal failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Seizure (General disorders) | 1 (1) | 0 (0)
Thoracic injury (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2014-10-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT02227446/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT02227446/SAP_001.pdf